CLINICAL TRIAL: NCT03087994
Title: The Influence of Obesity on Level of Depression and Cognitive and Executive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: rmc027816ctil
Record Dates: First submitted 2017-03-06; First posted 2017-03-23 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- girls with obesity attending a dietary intervention (Experimental): Participants in this group will attend 12 meetings of dietary interventions that will be guided by a dietician.
  Interventions: Behavioral: Nutritional guidance intervention
- girls with obesity (Active Comparator): participants in this group will only receive nutrition guidance once during the study
  Interventions: Behavioral: Nutritional guidance intervention
- girls with normal weight (Active Comparator): participants in this group will only receive nutrition guidance once during the study
  Interventions: Behavioral: Nutritional guidance intervention

INTERVENTIONS:
Behavioral: Nutritional guidance intervention — participants in this group will attend 12 meeting of nutritional guidance
  Arms: girls with obesity attending a dietary intervention
Behavioral: Nutritional guidance intervention — Participants in this group will only receive nutrition guidance once during the study
  Arms: girls with normal weight; girls with obesity

SUMMARY:
The proposed study is a randomized, open, comparative research involving an intervention group and two control groups.

The aims of the study are: 1.To compare levels of depression in female adolescents with obesity and a control group of female adolescents with appropriate weight and height. 2. To investigate whether a decrease in weight due to a short range intervention program provided by dietician for female adolescents with obesity will lead to change in the levels of symptoms of depression and cognitive and executive functions in comparison to a control group of adolescent girls with obesity, matched in age that does not receive such an intervention program.

60 Female adolescents with obesity will be recruited to the study and will be randomized to 1 of two groups- 1. intervention group- participants in this group will attend an intervention program consisting of 12 meetings with dietician and will attend two study visits at the clinic- in the beginning of the study and after three months. 2.Control group- Participants in this group will only come to two study visits at the clinic. In the first two visits they will meet with a dietician and will receive nutrition guidance.

Another 30 girls with appropriate weight will be recruited to second control group- this group will come to two study visits at the clinic- in the beginning of the study and after three months. In the first visit participants will receive nutrition guidance by the dietician.

In the study visits the following procedures will be performed for all study groups: Blood tests, completion of psychological and nutritional questionnaires, completion of computerized tests and measurements of height, weight, fat mass and circumference of hips.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescent girls aged 12-17, who attend the Endocrinology Institute in Schneider Hospital and comply with the research criteria: obesity (BMI above percentile 85) and appropriate weight (BMI between percentiles 5-85).
2. Adolescent level according to Tanner: 4-5.
3. Participants with obesity: BMI above percentile 85 for age group.
4. Participants in control group with appropriate weight: BMI percentile 5-85 for age group.
5. Appropriate height (Percentiles 3-97 according to the CDC curve).
6. Parents' signature on informed consent form.

Exclusion Criteria:

1. Chronic illness or chronic use of medications.
2. Inability to comply with the research conditions.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
Psychological questionnaires | change from baseline Psychological questionnaires at 3 months and at 1 year
Nutritional questionnaires | change from baseline Nutritional questionnaires at 3 months and at 1 year

SECONDARY OUTCOMES:
height | change from baseline height at 3 months and at 1 year
weight | change from baseline weight at 3 months and at 1 year
fat mass | change from baseline fat mass at 3 months and at 1 year
circumference of hips | change from baseline circumference of hips at 3 months and at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Joseph MD Meirovitch, Prof., Principal Investigator — Schneider children Medical center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No